CLINICAL TRIAL: NCT02020642
Title: Prospective Interventional Study Investigating the Effect of Renal Transplantation on Obstructive Sleep Apnea and Its Correlation to Nocturnal Rostral Fluid Shift, in End Stage Renal Disease Patients
Brief Title: Effect of Renal Transplantation on Obstructive Sleep Apnea in End Stage Renal Disease Patients (SASinTx)
Acronym: SASinTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Adam Ogna, Centre d'Investigation et Recherche sur le Sommeil (CIRS), Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIRS-SASinTx
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Obstructive Sleep Apnea; Overhydration; End Stage Renal Disease; Renal Transplantation
Keywords: polysomnography; bioimpedance; leg fluid shift; neck circumference; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Disorders, Intrinsic; Sleep Disorders; Apnea; Kidney Diseases; Kidney Failure, Chronic; Renal Insufficiency, Chronic; Renal Insufficiency; Dyssomnias
MeSH Terms: conditions — Sleep Apnea, Obstructive; Water Intoxication; Kidney Failure, Chronic; Sleep Apnea Syndromes; Sleep Disorders, Intrinsic; Sleep Wake Disorders; Apnea; Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency; Dyssomnias | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): A baseline polysomnography (PSG) is performed at inclusion (before renal transplantation, Tx), followed by a post-Tx PSG 6 months after transplantation
  Interventions: Procedure: Renal transplantation
- Control Group (No Intervention): A baseline polysomnography (PSG) is performed at inclusion, followed by a follow-up PSG at 6 months if the patient is not already transplanted

INTERVENTIONS:
Procedure: Renal transplantation — Renal transplantation from cadaveric or live donor
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to investigate the effect of renal transplantation on fluid overload and its consequence on the severity of obstructive sleep apnea, in patients with end stage chronic kidney disease. It aims further to investigate the relationship between overhydration, nocturnal rostral fluid shift and the severity of sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep disordered breathing is more prevalent in end stage kidney disease patients than in the general population, and may participate to the increased cardiovascular mortality observed in this group of patients. Despite a significant increase in knowledge about the harmful effects of obstructive sleep apnea, the pathophysiological mechanisms are poorly understood. Recent observations suggest a causative relationship between overnight fluid displacement from the legs to the neck soft and the severity of obstructive sleep apnea. This mechanism was demonstrated in otherwise healthy subjects, in heart failure patients, and in patients with venous insufficiency. We thus suspect that this pathophysiologic mechanism could explain the increased prevalence of obstructive sleep apnea in patients with fluid overload, including chronic renal failure.

The purpose of this study is to investigate the effect of renal transplantation on fluid overload and its consequence on the severity of obstructive sleep apnea, in patients with end stage chronic kidney disease. It aims further to investigate the relationship between overhydration, nocturnal rostral fluid shift and the severity of sleep apnea.

The severity of obstructive sleep apnea is measured by two attended polysomnographies, a baseline PSG performed before and a follow-up PSG performed 6 month after renal transplantation. Overhydration and leg fluid are evaluated by bioimpedance, performed at the beginning and at the end of each polysomnography. Patients who are not already transplanted 6 months after the baseline PSG will be re-assessed and will be analyzed as control group.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe obstructive sleep apnea, with an apnea-hypopnea index (AHI) ≥ 15/h
* age ≥ 18 years
* patient with end stage renal disease on waiting list for a renal transplantation (cadaveric or live donor).

Exclusion Criteria:

* unstable congestive heart failure
* active psychiatric disease
* amputation of the lower limbs, proximal to the ankle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Reduction of the obstructive sleep apnea severity | six months after renal transplantation
  Reduction of the obstructive sleep apnea severity, measured by attended polysomnography, six months after renal transplantation

SECONDARY OUTCOMES:
Reduction in nocturnal leg fluid volume shift between the legs and the neck | six months after renal transplantation
  Reduction in nocturnal leg fluid volume shift between the legs and the neck, measured by bioimpedance and neck circumference six months after renal transplantation
Relationship between overhydration, leg fluid volume shift, ankle and neck circumference and the severity of obstructive sleep apnea | at baseline and six months after renal transplantation
  Relationship between overhydration (measured by bioimpedance), leg fluid volume shift, ankle and neck circumference and the severity of obstructive sleep apnea
Change in the severity of the periodic limb movement disorder (PLMD) | six months after renal transplantation
  Change in the severity of the periodic limb movement disorder (PLMD)
Change in the severity of central sleep apnea | six months after renal transplantation
  Change in the severity of central sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Rapahël Heinzer, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV); Adam Ogna, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV); Valentina Forni Ogna, MD, Principal Investigator — Service de Néphrologie et Hypertension - Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (1):
- Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Forni Ogna V, Ogna A, Haba-Rubio J, Nowak G, Venetz JP, Golshayan D, Matter M, Burnier M, Pascual M, Heinzer R. Impact of kidney transplantation on sleep apnea severity: A prospective polysomnographic study. Am J Transplant. 2020 Jun;20(6):1659-1667. doi: 10.1111/ajt.15771. Epub 2020 Jan 21. PMID 31912961